CLINICAL TRIAL: NCT01771666
Title: A Pilot Study to Assess the Utility of Indocyanine Green™ (IC-GREEN™) SPY Imaging in the Mapping of Arm Draining Lymphatics and Nodes During Sentinel Node Resection With or Without Axillary Dissection in Breast Cancer
Brief Title: Pilot Indocyanine Green Imaging for Mapping of Arm Draining Lymphatics & Nodes in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Irene L. Wapnir, Professor - Med Center Line, Surgery - General Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-21030; SU-06122012-10130 (Other: Stanford University); BRS0022 (Other: OnCore)
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ISB and ICG (Experimental): The dose of Isosulfan blue (ISB) dye and Indocyanine green (ICG) solution will be started.
  (IC-GREEN) SPY Elite Imaging willbe used to capture the images of axillary cavity.
  Interventions: Device: SPY Elite Imaging; Drug: Indocyanine Green; Drug: Isosulfan blue; Drug: 99technetium-sulfur colloid radiolabel

INTERVENTIONS:
Device: SPY Elite Imaging — A camera that is directed into the axillary cavity to try to capture an image of the tumor site labeled with Indocyanine green before and after excising sentinel nodes
Drug: Indocyanine Green — started at 1mg /mL
  If fluorescence is not detected with this dose, then it will be increased by 50%.
  Other Names: IC-GREEN; ICG
Drug: Isosulfan blue — 3 to 5 mL
  If fluorescence is not detected with this dose, then it will be increased by 50%.
  Other Names: IS-BLUE; ISB; Lymphazurin
Drug: 99technetium-sulfur colloid radiolabel
  Other Names: 99tech

SUMMARY:
The purpose of this study is to determine if Indocyanine Green (IC-GREEN) is comparable to isosulfan blue (IS-BLUE) in the identification of arm lymphatics and arm-draining nodes during nodal staging procedures in breast cancer.

DETAILED DESCRIPTION:
It is the objective of the current study to test Indocyanine Green (IC-GREEN) as an agent for mapping arm draining lymphatics and nodes and compare it to isosulfan blue (IS-BLUE) in the setting of sentinel node procedures with or without axillary node dissections in women with breast cancer. All participants will also have tumor samples evaluated with 99technetium-sulfur colloid, a radiolabel used to identify tumor markers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Signed written informed consent.
* Women undergoing sentinel lymph node biopsy.
* Women with breast cancer with known or suspected lymph node involvement.
* Women undergoing sentinel node identification and completion axillary lymph node dissection.
* Women of 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) or Karnofsky Performance Status 0,1,2.
* Complete Blood Count (CBC) and basic Metabolic Panel within 6 months

Exclusion Criteria:

* History of liver or kidney failure will not be eligible.
* Allergies to iodine containing products will not be eligible.
* Women who are pregnant will not be eligible.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03-17 (Actual); Study Completion 2015-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Wapnir, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ISB and IC-Green Dye: The dose of Isosulfan blue (ISB) dye is 3 to 5 mL and Indocyanine green solution will be started at 1 mg/mL. If fluorescence is not detected with this dose, then it will be increased by 50%. A gamma probe [Neoprobe 2010] will be used to localize the sentinel lymph nodes in the axilla.
Period: Overall Study
Arm/Group | ISB and IC-Green Dye
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ISB and IC-Green Dye
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Agreement of Labeling Between Isosulfan Blue (IS-BLUE) and Indocyanine Green (IC-GREEN)
Description: Number of women with agreement of the two dies [ie, isosulfan blue (IS-BLUE) and indocyanine green (IC-GREEN)] on all nodes examined in the lymphatics and arm-draining lymph nodes, during nodal staging procedures for surgery to treat breast cancer with curative intent.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | ISB and IC-Green Dye
Number analyzed (Participants) | 23
Participants | 8

2. Secondary Outcome: Detection of Indocyanine Green (IC-GREEN); Isosulfan Blue (IS-BLUE); and 99technetium-sulfur Colloid Radiolabel in Resected Sentinel Nodes
Description: The outcome is expressed as the number of participants whose resected sentinel lymph nodes (SLN) bound 99technetium-sulfur colloid (99tech), a tumor marker radiolabel; Indocyanine Green (IC-GREEN; "GREEN"), a fluorescent label; or isosulfan blue (IS-BLUE; "BLUE"), a visual dye. Results are expressed as:
  * "Any HOT" = Those whose samples bound 99tech.
  * "Not HOT" = Those whose samples did not bind 99tech.
  * "Not HOT (also no BLUE, no GREEN)" = Those whose samples did not bind 99tech; and also did not bind IC-GREEN nor IS-BLUE.
  * "HOT, BLUE, GREEN" = Those whose samples bound all of 99tech; IC-GREEN; and IS-BLUE.
  * "HOT, no BLUE, no GREEN" = Those whose samples bound 99tech, but did not bind either of IC-GREEN nor IS-BLUE.
  * "HOT, GREEN only, no BLUE" = Those whose samples bound 99tech and IC-GREEN, but did not bind IS-BLUE.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | ISB and IC-Green Dye
Number analyzed (Participants) | 23
participants
  Any HOT | 20
  Not HOT (also no BLUE, no GREEN) | 3
  HOT, no BLUE, no GREEN | 12
  HOT, BLUE, GREEN | 6
  HOT, GREEN only, no BLUE | 2

ADVERSE EVENTS:
Arm/Group | ISB and IC-Green Dye
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes